CLINICAL TRIAL: NCT00128453
Title: Treatment and Prevention of Pericarditis With Colchicine. A Multicenter Double Blind Randomized Trial. The ICAP Trial: Investigation on Colchicine for Acute Pericarditis
Brief Title: Study of Colchicine to Treat Acute Pericarditis and Prevent Recurrences
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Sanitaria Locale 3, Torino (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCASL30501-1; EUDRACT number 2005-001570-28
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Pericarditis
Keywords: Pericarditis; Recurrence; Therapeutics; Prevention; Colchicine
MeSH Terms: conditions — Pericarditis; Recurrence | interventions — Colchicine; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Conventional therapy plus placebo
  Interventions: Drug: Placebo
- Colchicine (Active Comparator): Conventional therapy plus colchicine
  Interventions: Drug: Colchicine (for 3 months)

INTERVENTIONS:
Drug: Colchicine (for 3 months) — Colchicine 0.5mg BID (patients>70Kg) or 0.5mg once daily
  Arms: Colchicine
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether colchicine is safe and effective in the treatment of acute pericarditis and the prevention of subsequent recurrences.

DETAILED DESCRIPTION:
Colchicine is safe and effective in the management of recurrent pericarditis after failure of conventional treatment. Preliminary data have shown that it may be effective also in treatment of the index attack of pericarditis and the prevention of further recurrences.

Comparisons: The study will compare the safety and efficacy of colchicine in the treatment of acute pericarditis and the primary prevention of recurrences. Colchicine will be used in addition to conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute pericarditis (index attack)
* Age≥ 18 years
* Informed consent

Exclusion Criteria:

* Suspected neoplastic, tuberculous, or purulent etiology
* Known severe liver disease and/or elevated transaminases >1.5 times the upper limit of normality
* Serum creatinine >2.5 mg/dl
* Serum creatine kinase (CK) over the upper limit of normality or known myopathy
* Known gastrointestinal or blood disease
* Pregnant or lactating women or women not protected by a contraception method
* Known hypersensibility to colchicine
* Treatment with colchicine at enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2005-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Recurrence rate at 18 months | 18 months

SECONDARY OUTCOMES:
Symptom persistence at 72 hours, remission rate at 1 week | 1 week
Number of recurrences | 18 months
Time to first recurrence | 18 months
Disease-related re-hospitalization, cardiac tamponade, constrictive pericarditis within the duration of the study | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Rita TRINCHERO, MD, Study Chair — Cardiology Department. Maria Vittoria Hospital, ASL 3 Torino. Italy.; Massimo IMAZIO, MD, Study Chair — Cardiology Department. Maria Vittoria Hospital, ASL 3 Torino. Italy.; Massimo IMAZIO, MD, Principal Investigator — Cardiology Department. Maria Vittoria Hospital, ASL 3 Torino. Italy.
Locations (4):
- Italy (4):
  - Cardiology Department. Maria Vittoria Hospital, ASL 3 Torino, Torino, Torino
  - Internal Medicine Division, Bergamo
  - Cardiology Department-Ospedale Regionale, Bolzano
  - Ospedale di Rivoli, Rivoli

REFERENCES:
- [Background] Imazio M, Cecchi E, Ierna S, Trinchero R; ICAP Investigators. Investigation on Colchicine for Acute Pericarditis: a multicenter randomized placebo-controlled trial evaluating the clinical benefits of colchicine as adjunct to conventional therapy in the treatment and prevention of pericarditis; study design amd rationale. J Cardiovasc Med (Hagerstown). 2007 Aug;8(8):613-7. doi: 10.2459/01.JCM.0000281702.46359.07. PMID 17667033
- [Derived] Imazio M, Brucato A, Cemin R, Ferrua S, Maggiolini S, Beqaraj F, Demarie D, Forno D, Ferro S, Maestroni S, Belli R, Trinchero R, Spodick DH, Adler Y; ICAP Investigators. A randomized trial of colchicine for acute pericarditis. N Engl J Med. 2013 Oct 17;369(16):1522-8. doi: 10.1056/NEJMoa1208536. Epub 2013 Aug 31. PMID 23992557